CLINICAL TRIAL: NCT02637505
Title: Focal Cartilage Defects in the Knee - A Randomized Controlled Trial Comparing Arthroscopic Microfracture With Arthroscopic Debridement
Brief Title: Norwegian Cartilage Project - Microfracture
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University Hospital, Akershus (Other)
Collaborators: Kristiansund Hospital (Other); Alesund Hospital (Other); Haukeland University Hospital (Other); Diakonhjemmet Hospital (Other); Oslo University Hospital (Other); Haraldsplass Deaconess Hospital (Other)
Responsible Party: Principal Investigator, Asbjorn Aroen, Professor, University Hospital, Akershus
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2015/2202
Record Dates: First submitted 2015-12-15; First posted 2015-12-22 (Estimated); Last update posted 2025-01-07 (Actual); Status verified 2025-01

CONDITIONS: Knee Injury; Cartilage Injury
Keywords: Articular cartilage; Focal cartilage injury; Focal cartilage injury in the knee; Knee cartilage; Microfracture; Debridement
MeSH Terms: conditions — Knee Injuries; Fractures, Stress | interventions — Arthroplasty, Subchondral

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arthroscopic microfracture (MF) (Active Comparator): The AM group will be subjected to a diagnostic arthroscopy with a full inspection of the knee joint to ensure the inclusion criteria are fulfilled. The cartilage is cut sharp forming a rim of 90 degrees. The calcified layer is removed using a curette before an arthroscopic awl is then used to perform multiple holes ("microfractures") from the periphery towards the center. The microfractures are 3 - 4 mm apart and 2 - 4 mm deep into the subchondral bone. The correct and successful technique is confirmed by direct visualization: while reducing the fluid pump pressure, the release of marrow fat droplets and blood will be observed.
  Interventions: Procedure: Arthroscopic microfracture (MF)
- Arthroscopic debridement (AD) (Sham Comparator): The AD group will be subjected to a diagnostic arthroscopy with a full inspection of the knee joint to ensure the inclusion criteria are fulfilled. The lesion is stabilized, debriding all loose or marginally attached cartilage from the surrounding rim to form a stable edge of healthy cartilage around the defect using a ring curette, where cartilage slops down to the defect.
  Interventions: Procedure: Arthroscopic debridement (AD)

INTERVENTIONS:
Procedure: Arthroscopic microfracture (MF) — Arthroscopy With microfracture procedure
  Arms: Arthroscopic microfracture (MF)
Procedure: Arthroscopic debridement (AD) — Arthroscopy With debridement procedure
  Arms: Arthroscopic debridement (AD)

SUMMARY:
114 patients between 18 and 50 years with an isolated focal cartilage defect in the knee will be randomized to either receive arthroscopic microfracture or arthroscopic debridement. Both groups will then undergo a systematic physiotherapy training regime for 6-9 months. The groups will then be compared for results, after 3, 6, 12 and 24 months, by using validated patient reported outcome scores (Lysholm, KOOS, Tegner) and EQ5D as well as clinical examination and radiological findings at 2 years (MRI).

DETAILED DESCRIPTION:
Focal cartilage defects in the knee - A randomized controlled trial comparing arthroscopic microfracture with arthroscopic debridement.

Clinical compare the effect of arthroscopic microfracture (MF) with arthroscopic debridement (AD) in patients with symptomatic full thickness knee cartilage injuries less than 2cm2.

Focal cartilage injuries in the knee might have devastating effect both in the short term and in the long term. Various surgical treatment options are available, with microfracture the most used technique globally. Meta-analysis and systematic reviews have required well-designed, long-term, multicenter studies to evaluate clinical outcomes of microfracture with the use of a "no treatment" group as a control group.

H0: There is no difference in KOOS QoL after AM or AD 24 months after surgery. H1: There is a difference in KOOS QoL after AM or AD 24 months after surgery.

Questionnaires: KOOS, Tegner score, Lysholm score, EQ-5D, VAS. Physical examination: range of motion and hop test. Radiology: x-ray and MRI of the knee.

Primary aim: KOOS quality of life (QoL) subscore.

Prospective, double-blinded parallel-group multicenter study with 2 treatment arms. Approx. 24 months inclusion and 24 months follow up. In total 4 years.

All will be invited to participate in late controls after 5 and 10 years.

6 Norwegian hospitals: Akershus University Hospital, Oslo University Hospital - Ullevaal, Kristiansund Hospital, Aalesund Hospital, Diakonhjemmet Hospital and Haukeland University Hospital.

114 patients Inclusion: age 18-50 years old, single symptomatic cartilage defect on femoral condyle or trochlea.

2 treatment groups with 57 patients in each group. Follow up after 3 months (± 2 weeks), 6 months (± 4 weeks), 12 months (± 6 weeks) and 24 months (± 8 weeks). All will be invited to participate in late controls after 5 and 10 years. If any unforeseen complication outside normal clinical practice occurs, the sponsor representative will be contacted as soon as possible with a parallel message to the local coordinators at the involved hospitals. During each follow up, there will be a case report form (CRF) regarding complications and safety.

A 5 mL venous blood sample will be drawn on the day of operation. The blood sample will be centrifuged before serum is pipetted in a sterile tube. The serum will be analyzed at Oslo University Hospital - Rikshospitalet on the cartilage biomarker microRNA-140 (miR-140).

If normal distribution, aims will be analyzed using linear mixed models (LMM), and the primary aim will be performed as a post hoc test for the LMM, similar to performing a two-sample t-test. If no normal distribution, analysis will be performed using Mann-Whitney U-test.

Detecting a difference of 10 with 80 percent Power, uing a standard deviation of 18, this yields 52 patients in each group. By adding 10% due to loss during follow-up, we therefore plan to include a total of 114 patients.

No interim analysis will be done. Monitor from Health Møre and Romsdal HF. The end of this study is 24 months after the last included patient.

ELIGIBILITY:
Inclusion Criteria:

* Single symptomatic lesion of the trochlea, medial or lateral femoral condyle of the knee less than 2 cm2
* Cartilage lesion ICRS grade 3 or 4
* More than 50 % of the menisci intact
* Ligamentous stable knee
* Lysholm Score < 75
* Acceptable range of motion (5-105 degrees)

Exclusion Criteria:

* Osteoarthritis
* Malalignment > 5 degrees measured clinically, and if uncertainty on HKA radiographs
* Systemic arthritis
* Previous cartilage surgery except OCD fixation
* Obesity BMI > 30
* Serious drig or alcohol abuse
* Inability to answer questionnaires or partake in rehabilitation
* Comorbidity that may influence surgery or rehabilitation
* Pregnancy

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 66 (Actual)
Dates: Start 2016-01; Primary Completion 2024-12-31 (Actual); Study Completion 2024-12-31 (Actual)

PRIMARY OUTCOMES:
Knee Injury and Osteoarthritis Outcome Score (KOOS) Quality of Life | 24 months follow up
  The KOOS is a validated patient oriented outcome measure validated to use in cartilage Research. It assesses five domains, and the Fifth domain (knee related quality of life) will be the primary endpoint in this study. The primary aim is where the primary aim is the difference in KOOS QoL subscore in the AM group compared to the AD group at 24 months follow up.
  It is not planned any interim analysis before 24 months follow up.

SECONDARY OUTCOMES:
The Knee Injury and Osteoarthritis Outcome Score (KOOS) Other domains | 24 months follow up
  The other four domains of the KOOS score (pain, symptoms, Activity of daily living, sport and recreational function) will act as secondary endpoints
Tegner Score | 24 months follow up
  A validated knee-score to assess the level of physical Activity.
Lysholm Knee Score | 24 months follow up
  A condition specific knee score that assesses 8 domains: limp, locking, swelling, pain, stair climbing, use of support, instability and squatting.
EQ5D | 24 months follow up
  A generic measure of health status that produces a simple descriptive profile of Health status used in clinical evaluation of Health care.
Visual Analog Scale | 24 months follow up
  A visual analogue scale for pain, where 0 represents no pain and 10 represents the worst pain imaginable.
Range of motion | 24 months follow up
  Clinical evaluation of the joint range of motion
Magnetic Resonance Imaging (MRI) of the cartilage defect | 24 months follow up
  A radiographic evaluation (MRI) of the cartilage injury at 2 years, to evaluate which patients have adequate cartilage quality 2 years after surgery. The MRI will be taken with a cartilage specific protocol.
A Hop test | 24 months follow up
  Clinical evaluation of the knees agility, validated in knee sport medicine Research.

CONTACTS AND LOCATIONS:
Overall Officials: Tommy F Aae, MD,PhD, Principal Investigator — National coordinator; Øystein Lian, MD, Study Director — Kristian sund sykehus
Locations (1):
- Akershus University Hospital, Lørenskog, Norway

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Banitalebi H, Owesen C, Aroen A, Tran HT, Myklebust TA, Randsborg PH. Is T2 mapping reliable in evaluation of native and repair cartilage tissue of the knee? J Exp Orthop. 2021 Apr 28;8(1):34. doi: 10.1186/s40634-021-00350-1. PMID 33913035
- [Derived] Aae TF, Randsborg PH, Breen AB, Visnes H, Vindfeld S, Sivertsen EA, Loken S, Brinchmann J, Hanvold HA, Aroen A. Norwegican Cartilage Project - a study protocol for a double-blinded randomized controlled trial comparing arthroscopic microfracture with arthroscopic debridement in focal cartilage defects in the knee. BMC Musculoskelet Disord. 2016 Jul 16;17:292. doi: 10.1186/s12891-016-1156-y. PMID 27422025